CLINICAL TRIAL: NCT05178654
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE STUDY TO INVESTIGATE THE MASS BALANCE, METABOLISM AND EXCRETION OF [14C]PF-07321332 IN HEALTHY MALE PARTICIPANTS
Brief Title: Study to Investigate the Mass Balance, Metabolism, and Excretion of [14C]PF-07321332 in Healthy Male Participants.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on various healthy authorities feedback on PAXLOVID submission, this study is no longer required.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C4671007
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Healthy Participants
Keywords: Mass balance; metabolism and execration; COVID-19 (Coronavirus disease 2019); SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]PF-07321332 (Experimental): Single oral dose of 300 mg [14C]PF-07321332 containing approximately 100 µCi [14C]PF-07321332 coadministered with 100 mg ritonavir.
  Interventions: Drug: [14C]PF-07321332

INTERVENTIONS:
Drug: [14C]PF-07321332 — Single oral dose of 300 mg [14C]PF-07321332 containing approximately 100 µCi [14C]PF-07321332 coadministered with 100 mg ritonavir.

SUMMARY:
This study is to characterize mass balance and further the understanding of human pharmacokinetics, metabolism, and excretion of radiolabeled [14C]PF-07321332 in healthy male participants following oral administration with ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination (PE), laboratory tests, vital signs and standard 12 lead ECGs.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B surface antibody (HCVAb). Hepatitis B vaccination is allowed.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Participant who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.
* Participants enrolled in a previous radio-nucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry (ie, occupational exposure of 5 rems per year).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative amount of radioactivity Recovered in Urine (Ae) | 0 to 240 hours
  Ae is the cumulative amount of radioactivity recovered in urine. Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval. Sample volume = (urine weight in gram [g]/1.020), where 1.020 g/mL is the approximate specific gravity of urine.
Cumulative amount of radioactivity Recovered in Feces (Ae) | 0 to 240 hours
  Fe is the cumulative amount of radioactivity recovered in feces. Cumulative amount was calculated as sum of feces drug concentration in sample volume for each collection interval. Sample volume = (feces weight in gram [g]).
Metabolic Profiling in blood | 0 to 24 hours
  Metabolic profiling/identification and determination of relative abundance of [14C]PF-07321332 and the metabolites of [14C]PF-07321332 in plasma if possible.
Metabolic Profiling in Urine | 0 to 240 hours
  Metabolic profiling/identification and determination of relative abundance of [14C]PF-07321332 and the metabolites of [14C]PF-07321332 in urine if possible.
Metabolic Profiling in Feces | 0 to 240 hours
  Metabolic profiling/identification and determination of relative abundance of [14C]PF-07321332 and the metabolites of [14C]PF-07321332 in feces if possible.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 28 days after last dose of study medication
Number of Participants With Notable Electrocardiogram (ECG) Values | From baseline up to 11 days.
Number of Participants With Clinically Notable Vital Signs | From baseline up to 11 days
Number of Participants With Clinically Notable Clinical Chemistry/Biochemistry Shifts Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade | From baseline up to 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671007